CLINICAL TRIAL: NCT07300319
Title: The Effects of Chiropractic Care on Adults With Chronic Cancer-related Fatigue: a Pilot Trial
Brief Title: The Effects of Chiropractic on Cancer-related Fatigue
Acronym: CAN
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Life University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: I-0037
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Cancer; Fatigue
Keywords: Cancer; Fatigue; Chiropractic Care; Delayed Start
MeSH Terms: conditions — Neoplasms; Fatigue

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed Group (Active Comparator): After the 6-week lab assessments, the participants in the delayed group will be offered 6 weeks of chiropractic care.
  Interventions: Other: Delayed Chiropractic Care
- Immediate Group (Experimental): After the baseline assessment, the participants in the intervention group will receive 12 weeks of chiropractic care.
  Interventions: Other: Immediate Chiropractic Care

INTERVENTIONS:
Other: Immediate Chiropractic Care — Participants in the immediate start group will be assigned to chiropractic care for 12 weeks. Participants will have their upper cervical spine (C1/C2) assessed for the presence of vertebral subluxations per the chiropractor's normal and customary procedures and adjusted if necessary.
  Arms: Immediate Group
Other: Delayed Chiropractic Care — Participants in the delayed start group will be assigned to chiropractic care for 6 weeks. Participants will have their upper cervical spine (C1/C2) assessed for the presence of vertebral subluxations per the chiropractor's normal and customary procedures and adjusted if necessary.
  Arms: Delayed Group

SUMMARY:
The goal of this randomized controlled study is to investigate the impact of chiropractic care on CCRF (Chronic Cancer Related Fatigue) and other health-related challenges that burden cancer survivors.

DETAILED DESCRIPTION:
To our knowledge, the impact of chiropractic care on CCRF and other health-related challenges that burden cancer survivors has yet to be investigated. Because this is a pilot trial, the primary outcomes center around feasibility and include 1) randomization, 2) compliance, 3) tolerability, 4) adherence, and 5) retention in each arm. Secondary outcomes include changes in patient-reported outcomes (PROs), electrocardiography (ECG) derived heart rate variability (HRV), impedance cardiography (ICG) derived pre-ejection period (PEP), and number of completed sit-to-stands.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age.
* Self-report that they have been informed by their primary health care provider that they are cancer-free (this is sometimes referred to as 'complete remission' or 'cured').
* Minimum of 3 months since the completion of their primary curative-intent cancer therapies including surgery, chemotherapy, radiotherapy, and/or immunotherapy (long-term hormone therapy permitted)
* Scores in the moderate-to-severe range (i.e., at or above the 60th percentile) on the FACIT-Fatigue scale.
* Fatigue onset was at some point during their illness/treatment & negatively impacts their quality of life & daily functioning.

Exclusion Criteria:

* Chiropractic care within the past 2 weeks
* Taking short-acting benzodiazepines which include midazolam/Versed & triazolam/Halcion.
* Taking GLP-1 medications
* Taking other types of prescription medications (including hormone therapy) and hasn't been on a stable dose for a minimum of 6 weeks with plans to change medications or doses during the study.
* Disorders that cause fainting during rapid postural changes (e.g., POTS, orthostatic hypotension).
* Not able to make a fist or grip objects with one or both hands
* Deaf in one or both ears (hearing aids are ok)
* Heart conditions, including pacemakers, which impact heart function
* Diagnosed with rheumatoid arthritis, osteoporosis, or medically diagnosed cervical spine instability.
* Current litigation related to a physical, health-related injury.
* Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of Eligible Randomized Participants | 2 years
  The proportion of eligible participants randomized into the study
Number of Participants Who Adhere to Study | 2 years
  Proportion of enrolled participants who adhere to the pre-baseline assessment lifestyle restrictions as instructed. This assesses compliance.
Number of Participants That Can Fulfill Study Activities | 2 years
  Proportion of participants that can fulfill the given baseline assessment as directed. This assesses tolerability
Number of Participants Who Chiropractic Sessions | 2 years
  Proportion of randomized adults attending ≥90% of chiro sessions within 7 days of the prescribed time frame. This assesses adherence to treatment.
Number of Enrolled Intervention Group Participants | 2 years
  Proportion of the immediate-start group attending the final assessment session. This assesses retention.

CONTACTS AND LOCATIONS:
Overall Officials: Tyson Perez, DC, PhD, Principal Investigator — Life University
Locations (1):
- Center for Chiropractic Research, Marietta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No